CLINICAL TRIAL: NCT05305547
Title: A Phase 3, Multicenter, Randomized, Double-Blind, 24-Week Study of the Clinical and Antiviral Effect of S-217622 Compared With Placebo in Non-Hospitalized Participants With COVID-19
Brief Title: A Study to Compare S-217622 With Placebo in Non-Hospitalized Participants With COVID-19
Acronym: SCORPIO-HR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTIV-2d/A5407
Record Dates: First submitted 2022-03-30; First posted 2022-03-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — ensitrelvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S-217622 (Experimental): S-217622 will be administered orally for 5 days.
  Interventions: Drug: S-217622
- Placebo (Placebo Comparator): Placebo matching to S-217622 will be administered orally for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-217622 — Administered as a round tablet.
  Arms: S-217622
Drug: Placebo — Administered as a round tablet.
  Arms: Placebo

SUMMARY:
The main aim of this study is to evaluate the efficacy of S-217622 versus placebo among outpatient adults with mild and moderate COVID-19 starting intervention within 3 days of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of laboratory-confirmed active SARS-CoV-2 infection, as determined by a nucleic acid (for example, reverse-transcriptase PCR) or antigen test from any respiratory tract specimen (for example, oropharyngeal, NP or nasal swab, or saliva) collected ≤72 hours (3 days) prior to randomization.
* Participants are expected to begin study intervention ≤3 days from self-reported date of onset of any of the COVID-19-related symptoms from the following list:
* Cough
* Shortness of breath or difficulty breathing
* Feeling feverish
* Chills
* Fatigue
* Body pain or muscle pain or aches
* Diarrhea
* Nausea
* Vomiting
* Headache
* Sore throat
* Nasal obstruction or congestion
* Nasal discharge
* Loss of taste
* Loss of smell
* One or more of the following signs/symptoms present within 24 hours prior to randomization:
* Cough
* Shortness of breath or difficulty breathing
* Feeling feverish
* Chills
* Fatigue
* Body pain or muscle pain or aches
* Diarrhea
* Nausea
* Vomiting
* Headache
* Sore throat
* Nasal obstruction or congestion
* Nasal discharge
* Participants at higher risk of progression to severe COVID-19 are defined as follows:
* Age ≥65 years
* Age ≥18 with 1 of the following:
* Obesity (body mass index [BMI] ≥30 kilograms per square meter [kg/m^2]). Note: BMI is rounded to the nearest whole number, for example 29.5 kg/m^2 is rounded to 30 kg/m^2.
* Diabetes mellitus
* Hypertension requiring daily prescribed therapy
* Cardiovascular disease (requiring daily prescribed therapy or congenital heart disease)
* Chronic lung disease (for example, chronic obstructive pulmonary disease, moderate to severe asthma, interstitial lung disease, cystic fibrosis, pulmonary hypertension) requiring daily prescribed therapy
* Chronic kidney disease, defined as known current kidney impairment with a creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) <60 milliliters (mL)/minute (min)/1.73 square meter (m^2) within the past 12 months prior to randomization, as long as the participant does not have known CrCl <30 mL/min by Cockcroft-Gault or require dialysis
* Down syndrome
* Sickle cell disease
* One of the following immunocompromising conditions or immunosuppressive treatments:
* Receiving chemotherapy or other therapies for cancer
* Hematologic malignancy (active or in remission)
* History of a hematopoietic stem cell or a solid organ transplant
* Human immunodeficiency virus infection: not on antiretroviral therapy or with cluster of differentiation 4+ cell count <200 cells per cubic millimeter
* Combined primary immunodeficiency disorder
* Taking immunosuppressive medications (for example, drugs to suppress rejection of transplanted organs or to treat rheumatologic and gastrointestinal conditions, such as anti-tumor necrosis factor agents, mycophenolate, and rituximab).

Note: Current use of some corticosteroids is exclusionary, due to concern for possible drug-drug interaction (DDI) with S-217622.

Exclusion Criteria:

* History of hospitalization for the current SARS-CoV-2 infection (that is, prior hospitalization for a prior episode of SARS-CoV-2 infection is allowable)
* For the current SARS-CoV-2 infection, any positive SARS-CoV-2 molecular (nucleic acid) or antigen test from any respiratory tract specimen (for example, oropharyngeal, NP, or nasal swab, or saliva) collected ˃72 hours (3 days) prior to randomization. Participants with reinfection, defined as prior SARS-CoV-2 infection that began >90 days prior to the current onset of symptoms with interval resolution of symptoms are eligible as long as the current infection has not been present for more than 3 days prior to randomization.
* Current need for hospitalization or immediate medical attention in the opinion of the investigator
* Current use of any medications prohibited with the study intervention. Individuals who have used Paxlovid or any other oral, inhaled, or injectable medication intended to treat the current SARS-CoV-2 infection before randomization are excluded. After randomization, locally available SARS-CoV-2 treatment (including but not limited to molnupiravir, mAbs, outpatient IV remdesivir, convalescent plasma, inhaled budesonide, favipiravir, and fluvoxamine) will be permitted, as long as there are no concerns for DDIs.

Note: Paxlovid use for a prior episode of COVID-19 is permitted.

* Receipt of any investigational treatments for the current episode of SARS-CoV-2 at any time prior to randomization is exclusionary. Note: This does not include drugs approved for other uses and taken for those indications or COVID-19 vaccines. Note: Use of locally authorized or approved therapies to prevent COVID-19, such as mAbs given solely to prevent COVID-19, are not exclusionary.
* Any co-morbidity requiring surgery within 7 days prior to randomization or that is considered life threatening in the opinion of the investigator within 28 days prior to randomization
* Known allergy/sensitivity or any hypersensitivity to components of S-217622 or placebo for S-217622
* Known (within 12 months prior to randomization) renal impairment defined as CrCl <30 mL/min by Cockcroft-Gault or requiring dialysis
* Known history of cirrhosis or liver decompensation (including ascites, variceal bleeding, or hepatic encephalopathy)
* Participants who have used any of the following drugs within 14 days prior to randomization:
* Strong cytochrome P453A inducer
* Products containing St. John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2093 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Median Time to Sustained Symptom Resolution | Up to Day 29

SECONDARY OUTCOMES:
Change From Baseline in Quantitative log10 SARS-CoV-2 RNA Levels by Polymerase Chain Reaction (PCR) on Nasopharyngeal (NP) Swab at Day 4 | Baseline, Day 4
Percentage of Participants With Adjudicated Hospitalization Due to COVID-19 or Death Due to Any Cause | Up to Day 29
Percentage of Participants With Detectable SARS-CoV-2 by Viral Culture on NP Swab at Day 4 | Day 4
Percentage of Participants With Hospitalization (All Cause) or Death Due to Any Cause | Up to Day 29
Percentage of Participants With Detectable SARS-CoV-2 by Viral Culture on NP Swab at Day 8 | Day 8
Percentage of Participants With NP SARS-CoV-2 RNA Levels by Quantitative PCR Below the Lower Limit of Quantification on Days 4 and 8 | Days 4 and 8
Median Change From Baseline of SARS-CoV-2 RNA by Quantitative PCR in NP Swabs on Day 8 | Baseline, Day 8
Median Time to Self-Reported Return to Usual (Pre-COVID-19) Health | Up to Day 29
Percentage of Participants Reaching a Score ≥2, ≥3, ≥4, ≥5, ≥6, ≥7, or ≥8 on the Ordinal Scale | Up to Day 29
Change From Baseline in Resting Peripheral Oxygen Saturation at Day 29 | Baseline, Day 29
Percentage of Participants With Resting Peripheral Oxygen Saturation ≥96% | Up to Day 29
Percentage of Participants Exhibiting Persistent and/or Late-Onset Symptoms | Up to Weeks 12 and 24
Percentage of Participants With Symptomatic Viral Rebound as an Increase in Quantitative NP SARS-CoV-2 Viral Culture or NP SARS-CoV-2 RNA Levels by Quantitative PCR After Day 4 up to Day 29 | Day 4 up to Day 29
Percentage of Participants With Viral Rebound as an Increase in Quantitative NP SARS-CoV-2 Viral Culture or NP SARS-CoV-2 RNA Levels by Quantitative PCR After Day 4 up to Day 29 | Day 4 up to Day 29
Number of Participants With Adverse Events | Up to Week 24
Change From Baseline in Short Form 36 Version 2.0 (SF-36 V2) Quality of Life Score | Baseline, Week 24
Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score | Baseline, Week 24
Change From Baseline in Post-Acute COVID-19 Questionnaire | Baseline, Week 24
Percentage of Participants Who Experienced Death Due to Any Cause | Up to Week 24

CONTACTS AND LOCATIONS:
Locations (195):
- United States (53):
  - Lakeview Clinical Research, Guntersville, Alabama
  - Voyage Medical Services, Tempe, Arizona
  - Novak Clinical Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Carbon Health, Culver City, California
  - NICR, Garden Grove, California
  - Ark Clinical Research (PARENT), Long Beach, California
  - UCSD Antiviral Research Center, San Diego, California
  - University of California San Francisco (PARENT), San Francisco, California
  - Clinical Trials Management Services, 223 E. Thousand Oaks Blvd., Thousand Oaks, California
  - Lundquist Institute for BMI, UCLA Medical Center, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - University of Florida Clinical & Translational Science Institute, Gainesville, Florida
  - Universal Medical and Research Center, Miami, Florida
  - CCR Medical Center, Suite 201, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Quantum Clinical Trials, 333 Arthur Godfrey Road, Suite 202, suite 208, Miami Beach, Florida
  - Quality Research of South Florida, Miami Lakes, Florida
  - Accel Research Sites Network, Ormond Clinical Research Unit, 77 West Granada Boulevard, Ormond Beach, Florida
  - Clinical Research Center of Florida, 550 SW 3rd St.,, Suite #305, Pompano Beach, Florida
  - Invictus Clinical Research Group, LLC, Pompano Beach, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Masters of Clinical Research, Augusta, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Research Network America, Berwyn, Illinois
  - Rush University Infectious Diseases, Chicago, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Infusion Associates, Grand Rapids, Michigan
  - Revival Research Institute LLC, Troy, Michigan
  - Las Vegas Medical Research, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Columbia University Irving Medical Center Division of Infectious Diseases, New York, New York
  - NY Blood Center Project ACHIEVE, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Lapis Clinical Research - North State, Denver, North Carolina
  - Burke Primary Care, Morgantown, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - Ohio State University College of Medicine, Columbus, Ohio
  - Infectious Disease Clinical Trials Unit-University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - UPMC Eye Center - Eye and Ear Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Health-One Hundred Oaks, Nashville, Tennessee
  - Central Texas Medical Research, Austin, Texas
  - Care United Research, 375 North FM 548, suite 100, Forney, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - Trio Clinical Trials, LLC., Houston, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Clinical Research Partners LLC, Richmond, Virginia
- Argentina (15):
  - CINME Centro Investigaciones Metabolicas, Pres. Jose Evaristo Uriburu 754, Piso 3 dpto 12, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Sanatorio De La Trinidad, Mitre Bartolome Mitre, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano sede Central, Tte. Gral. Juan Domingo Perón 4190, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Privado de Medicina Familiar, Mindout Research, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro De Investigaciones, Mar del Plata, Buenos Aires
  - DIM Clínica Privada, Belgrano 136 - 5to piso, Ramos Mejía, Buenos Aires
  - Hospital General Agudos Dr. J.M., Grl Justo José de Urquiza 609 2do piso, Pabellón Clínica Médica, Enf. Emergentes, Ramos Mejía, Buenos Aires
  - Clínicas Zárate, F. Andrade 332, Zárate, Buenos Aires
  - Sanatorio Privado ,Duarte Quiros, Quiros, Córdoba Province
  - Instituto Médico de la, Fundación Estudios Clínicos, Italia 428, Rosario, Rosario, Sante Fe
  - Clinica Mayo UMCB, San Miguel de Tucumán, Tucumán Province
  - Clínica Olivos, Buenos Aires
  - Sanatorio Allende, Av., Córdoba
  - CER San Juan,, San Juan
  - Mendoza 2612, Rosario, Santa Fe
- Brazil (20):
  - SENAI CIMATEC Clinical Trial Research Center, Salvador, Estado de Bahia
  - AMB3 Servicos Medicos Ltda Rua Campinas, Cuiabá, Mato Grosso
  - Faculdade de Medicina da univ., Federal, Av Alfredo Balena, 190, 1° andar - sala 161, Belo Horizonte, Minas Gerais
  - Hosp Nossa Senhora das Gracas, Rue Alcides Munhoz, Curitiba, Paraná
  - Instituto Atena de Psequisa Clinica Ltds, Av Marechal Floriano Peixoto, Natal, Rio Grande do Norte
  - Thainá Garbino dos Santos, Avenida Protásio Alves 211, Bloco C, Porto Alegre, Rio Grande do Sul
  - IPARGS, Rua Antonio Joaquim Mesquita, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Amor de, Barretos; Rua Antenor Duarte Villela, Baretos, São Paulo
  - Unid Pesquisa Clínica Facultad Medicina, de Botucatu UNESP, Rua Prof. Dr. Armando,Alves s/n, Distrito de rubião Junior, Botucatu, São Paulo
  - Hospital Universario Sao Francisco, na Providencia de Deus-Av. Sao Francisco de Assis, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clinica de Campinas IPECC Tua Oswaldo, Campinas, São Paulo
  - Cecip Jau, Jaú, São Paulo
  - Pesquisare Saude, Santo André, São Paulo
  - CEMEC, São Bernardo do Campo, São Paulo
  - Esperanca Clinica De Pesquisas, São Paulo, São Paulo
  - Instituto de Molestast Cardiovasculares, Tatuí, São Paulo
  - Hospital da Puc Campinas, Centro de Pesquisa Sao Lucas, Campinas
  - IBPClin, Rua da Gloria, Rio de Janeiro
  - INI/Fiocruz, Rio de Janeiro
  - Lóbus Cntr. de Pesquisa Cl., Volta Redonda
- Colombia (9):
  - Programa de estudios y control de, enfermedades tropicales PECET, Carrera 53 N°61-30 Torre 2, Lab. 632, Medellín, Antioquia
  - Centro de Investigación Medico, Asistencia - CIMEDICAL S.A.S, Cra 49C # 82-120, Barranquilla, Atlántico
  - Corazon IPS S.A.S, Carrera 49 No 74 - 158, Barranquilla, Atlántico
  - IPS CENTRO CIENTIFICO ASISTENCIAL S.A.S, Cra 45 #85-49, Barranquilla, Atlántico
  - Centro de investigación en Reumatología, y Especialidades Medicas S.A.S, CIREEM S.A.S.-Cra. 12#97-32, Bogotá, Bogota D.C.
  - Fundación Centro Excelencia en Enferm., Crónicas No Transmisibles-FUNCENTRA, CRA 3 N°21 44 B,, Chuchurubi Monteria, Departamento de Córdoba
  - TyC Inversiones SAS Grupsalud 33-6 IPS, Avenida Libertador # 30-360, Barrio San Pedro Alejandrino, Santa Marta, Magdalena Department
  - Fundación Cardiomet Cequin,, Street 18 North # 14-25,, Armenia, Quindío Department
  - BlueCare Salud SAS, Bogotá
- Ghana (3):
  - Navrongo Health Research Cntr, Upper East, Navrongo
  - Kintampo Health Research Cntr, Kintampo
  - Kumasi Centre for Research, South End Asuogya Road, Kwame Nkrumah University, Kumasi
- India (26):
  - St. Theresa's Hospital, Hyderabad, Andhra Pradesh
  - DEC-Health Care Hospital, Nellore, Andhra Pradesh
  - Vijaya Super Speciality Hospital, Nellore, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Sangini Hospital 1st Flr & 7th flr, Ahmedabad, Gujarat
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Rhythm Heart Institute - A Unit Of SLPL, Vadodara, Gujarat
  - ESIC Medical College & Hospital, Faridabad, Haryana
  - Sarvodaya Hospital and Research Centre, Faridabad, Haryana
  - BGS Global institute of Medical Sciences, Bangalore, Karnataka
  - KLEs Dr. Prabhakar Kore Hospital & MRC Belagavi, Belagavi, Karnataka
  - Sri Lakshmi Super Speciality Hospital, Bengaluru, Karnataka
  - Shettys Hospital, Bengaluru, Karnataka
  - Sri Venkateshwara Hospitals, SKY HEIGHTS, Site#1/2, Sarjapura-Attibele, Main rd, Indelebele Village, Bengaluru, Karnataka
  - Yenepoya Med College Hosp, EMD Building, 5th fl., University Rd, Deralakatte, Mangalore, Karnataka
  - BAJ RR Hosp and Res Cntr, Dombivali, Maharashtra
  - Chopda Medicare & Research Centre Pvt. Ltd, Nashik, Maharashtra
  - Lifepoint Multispecialty Hosp., Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Aakash Healthcare Private Limited, Dwārka, New Delhi
  - JNUIMSRC, Jaipur, Rajasthan
  - Tagore Hospital & Research Institute, Jaipur, Rajasthan
  - Voluntary Health Services Infectious Diseases Medical CEN CART Clinical Research Site, Chennai, Tamil Nadu
  - Department of Medicine, Kanpur, Uttar Pradesh
  - HB Specialty Hosp. & Res Inst., Rudrapur, Uttarakhand
  - Calcutta School of Tropical Medicine, Kolkata, West Bengal
- Japan (5):
  - Kohokai Takagi Hospital, Okawa-shi, Fukuuoka-Ken
  - Tsuchiura Beryl Clinic, Tsuchiura-shi, Ibaraki
  - University of Tsukuba Hospital, Tsuchiura-shi, Ibaraki
  - Tashiro Endocrinology Clinic, Tsukuba, Ibaraki
  - Kodaira Hospital, Toda-shi, Saitama
- Kenya (2):
  - Moi University Clin Res Centre, 2nd Fl, Chandaria Chronic, Disease and Cancer Centre, Eldoret
  - KEMRI CGHR HIVR Site, Kisumu
- Malawi (3):
  - Johns Hopkins Research Project, Queen Elizabeth Central Hospital, Chipatala Avenue, Blantyre
  - UNC Project, Private Bag A-104, Lilongwe
  - Mangochi PHNG Study Site, Kamuzu University of Health Sciences, Private Bag 360, Room 805, Mangochi
- Mexico (8):
  - CAIMED Investigación en Salud, S.A. de C.V., Manzanillo #100. Piso 2. Roma Sur, Cuauhtémoc, Cdmx, C.P
  - Instituto Veracruzano, en Investigación Clínica S.C., Sabino s/n, Colonia Reserva Tarimoya ll, Veracruz, CP
  - Avenida Universidad 1001, Edificio 19, planta baja, colonia Chamilpa, Cuernavaca, Morelos
  - Oaxaca Site Management Organization S.C., Humboldt 302, Col. Centro., Oaxaca City, Oaxaca
  - Centro Inv. y Avances Med Especializados, (CIAME) Av. Kabah, Lote 38, 39 y 41., Manzana 4, supermanzana 44. Col., Alborada, Benito Juárez, Cancún, Quintana Roo
  - FAICIC S. DE R.L. DE C.V., Av. 16 de Septiembre 1165, Ricardo Flores Magón, Veracruz
  - Hospital Cardiológica Aguascalientes, Ecuador 200 Fracc Las Américas, Aguascalientes
  - Centro de Inv. Médica Aguascalientes, (CIMA) Av. Independencia 2130, Int. A. Trojes de Alonso, Aguascalientes
- Pakistan (10):
  - Indus Hospital and Health Network, Korangi, Karachi
  - Rehman Medical Institute Clinical Trial Unit, Hayatabad, Peshawar
  - Central Park Teaching Hospital, Lahore, Punjab Province
  - National Hospital & Medical Center, Lahore, Punjab Province
  - Akram Medical Complex, Lahore, Punjab Province
  - The Aga Khan University, Karachi, Sindh
  - Shifa International Hospital, 4 Pitras Bukhari Rd, H-8/4, H-8, Islamabad
  - Dow Univ of Health Sciences Ojha Campus, Karachi
  - Sindh Infectious Disease Hospital and research Centre, Karachi
  - Maroof International Hospital, Peshawar
- Peru (5):
  - Centro de Investigación, San Isidro, Lima region
  - Asoc. Civil Selva Amazonica, Iquitos, Loreto
  - Centro de Inv. Tecnológicas Biomédicas y Medioambientales, Lima
  - Asoc. Civil Impacta Salud y Educación - Sede San Miguel, Lima
  - Patricia Ortiz Bazan, Lima Cercado
- Philippines (8):
  - Mary Mediatrix Medical Cntr, Lipa, Batangas
  - Mary Johnston Hospital, 1221 Juan Nolasco Street, Tondo, Manila
  - Iloilo Doctors' Hospital, Room 706, New Condoclinics Bldg, West Ave, Lloilo, Molo
  - The Medical City Clark, #100Eatwick, Gatewick, Global Gateway Logistics City, Industrial Estate 5, Clark Freeport Zone, Mabalacat, Pampanga
  - Ilocos Training and Regional Medical Center, La Union, San Fernando
  - Green City Medical Center, Pampanga, San Fernando
  - Health Cube Medical Clinics, High Pointe Medical Hub, 241 Shaw Blvd, Mandaluyong
  - Lung Center of the Philippines, Quezon City
- Poland (5):
  - Ostrowieckie Centrum Medyczne, Ostrowiec Świętokrzyski
  - Medicome sp. z o.o., Oświęcim
  - Centrum Medyczne "Medyk", Rzeszów
  - Clinmedica Research sp. z o.o., Skierniewice
  - Centrum Badań Klinicznych, Wroclaw
- South Africa (15):
  - JOSHA Research, Bloemfontein, Free State
  - Newton Clinical Research Centre, Johanesburg, Gauteng
  - Worthwhile Clinical Trials, Johannesburg, Gauteng
  - (PHRU), New Nurses Home 9th floor Chris, Johannesburg, Gauteng
  - CHRU, Themba Lethu Clinic, Johannesburg, Gauteng
  - Ubuntu Clinical Research, Krugersdorp, Gauteng
  - Ubuntu Clinical Research, Lenasia, Gauteng
  - T/A Midrand Medical Centre, Shop #1, Health Emporium, Midrand, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - Right to Care Research Esizayo, Right Clinic Esizayo, Randburg, Gauteng
  - Limpopo Clin Res Initiative Tamboti Medical Centre, Thabazimbi, Limpopo
  - The Arum Institute NPC Rustenburg CRS, Rustenburg, North West
  - Task Eden Research Centre, George, Western Cape
  - Be Part Research PTY (LTD), Paarl, Western Cape
  - Roodepoort Medicross Clinical Research Centre, Roodepoort
- Thailand (4):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok
  - Srinagarind Hospital, Mueang Khon Kaen District, Changwat Khon Kaen
  - Research Institute for Health Sciences, Mueang Chiang Mai District, Chiang Mai
- Uganda (4):
  - Joint Clinical Research Centre, Kampala
  - Infectious Diseases Institute (IDI), Mulago Hill Road, Kampala
  - SICRA, Lira Regional Referral, Plot 21-41 Ngetta Road P.O. Box 330062, Lira
  - IDRC Clinic, Tororo General Hospital, P.O. Box 2, Station Rd, Tororo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luetkemeyer AF, Chew KW, Lacey S, Hughes MD, Harrison LJ, Daar ES, Eron J, Fletcher CV, Greninger AL, Hessinger D, Li JZ, Mailhot D, Wohl D, Chayakulkeeree M, Mendoza JLA, Elistratova P, Makinde O, Morgan G, Portsmouth S, Uehara T, Smith D, Currier JS. Ensitrelvir for the Treatment of Nonhospitalized Adults with COVID-19: Results from the SCORPIO-HR, Phase 3, Randomized, Double-blind, Placebo-Controlled Trial. Clin Infect Dis. 2025 Jul 18;80(6):1235-1244. doi: 10.1093/cid/ciaf029. PMID 39960062

DOCUMENTS (1):
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT05305547/ICF_000.pdf